CLINICAL TRIAL: NCT00215501
Title: A Phase I Trial of Capecitabine or Continuous Infusion 5-Fluorouracil in Combination With Weekly Irinotecan and Cisplatin in Patients With Advanced Solid Tumor Malignancies
Brief Title: Capecitabine or 5-Fluorouracil in Combination With Irinotecan and Cisplatin in Patients With Solid Tumor Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Peter C. Enzinger, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-042
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Solid Tumor
Keywords: advanced solid tumor malignancy; capecitabine; continuous infusion; 5-FU; irinotecan; 5-fluorouracil; cisplatin
MeSH Terms: interventions — Capecitabine; Fluorouracil; Irinotecan; Cisplatin

ARMS (2):
- Group A (Experimental): Oral capecitabine
  Interventions: Drug: Capecitabine; Drug: Irinotecan; Drug: Cisplatin
- Group B (Experimental): 5-fluorouracil
  Interventions: Drug: 5-Fluorouracil (5-FU); Drug: Irinotecan; Drug: Cisplatin

INTERVENTIONS:
Drug: Capecitabine — Orally twice a day for 14 days (dosage will vary)
  Arms: Group A
Drug: 5-Fluorouracil (5-FU) — Continuous infusion 24 hours a day for 14 days (Days 1-14) Dosage will vary
  Arms: Group B
Drug: Irinotecan — Intravenously weekly for 2 weeks (given after cisplatin) followed by a one-week rest period
Drug: Cisplatin — Intravenously weekly for 2 weeks followed by a one week rest period

SUMMARY:
The purpose of this study is to test the safety of irinotecan and cisplatin in combination with either capecitabine or continuous infusion 5-fluorouracil and to see what effects (good and bad) these have on patients with unresectable, advanced solid tumors.

DETAILED DESCRIPTION:
* This is a Phase I dose escalation study. The dose of drug the patient receives will be assigned based upon when they enter the study. Since we are looking for the highest dose of capecitabine or 5-fluorouracil that can be given safely in combination with cisplatin and irinotecan, not everyone who participates in this study will be receiving the same amount of the drug.
* There are four parts to this study: 1)Choice of treatment, 2)Evaluation, 3)Chemotherapy and 4)Follow-up.
* The patient and the patient's doctor will decide which form of chemotherapy is best for the patient, either pill form or continuous infusion. Chemotherapy pills (capecitabine) are given twice per day for 14 days is a row every 3 weeks. Continuous infusion (5-fluorouracil) is given through a pump 24 hours a day for 14 days every 3 weeks.
* Prior to initiation to therapy the extent of the patients cancer will be evaluated. This includes a CT scan, chest x-ray, EKG and bloodwork.
* Patient's will receive chemotherapy for 2 weeks followed by a one week break. This will constitute one cycle. The medications cisplatin and irinotecan will be given intravenously on the 1st and 8th day of each cycle. Following the rest period the next cycle of chemotherapy begins.
* Following 2 cycles of chemotherapy, the patients cancer will be re-evaluated. A CT scan and bloodwork will be obtained and will be compared to the previous studies. Treatment will resume if the cancer is the same size or smaller than before and the patient is tolerating the chemotherapy well. The cancer will be re-evaluated every 2 cycles of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor malignancy
* 18 years of age or older
* Two prior chemotherapy regimens for metastatic disease. Prior chemotherapy must have been completed at least 3 weeks prior to initiation of this protocol.
* ECOG performance status of 0,1 or 2
* Neutrophils greater or equal to 1,500/ul
* Platelets greater or equal to 100,000/ul
* Serum bilirubin less or equal to 1.5 mg/dl
* Creatinine clearance greater than 50 ml/min
* AST or SGOT less or equl to 3x ULN
* Prior radiotherapy is allowable, provided at least 4 weeks have elapsed and the patient has recovered from all therapy related side effects.

Exclusion Criteria:

* Life expectancy of less than 3 months
* Clinically significant cardiac disease or myocardial infarction within past 6 months
* Suspicion or documentation of CNS metastases or carcinomatous meningitis
* Psychiatric disability judged by the investigator to be clinically significant, precluding informed consent
* Known existing coagulopathy and/or requires therapeutic anticoagulants
* Uncontrolled diarrhea
* Peripheral neuropathy
* Major surgery within 3 weeks of the state of the study treatment without complete recovery
* Serious, uncontrolled, concurrent infection
* Lack of physical integrity of upper gastrointestinal tract or malabsorption syndrome
* Prior severe reaction to fluoropyrimidine, irinotecan or cisplatin
* Known interstitial pulmonary fibrosis
* Known Gilbert's disease
* Uncontrolled diabetes mellitus
* Organ allograft(s) on immunosuppressive therapy
* Pregnant or lactating women
* Patients taking valproic acid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2001-11; Primary Completion 2005-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To determine dose limiting toxicity, maximum tolerated dose and recommended Phase II dose of both capecitabine and 5-fluorouracil in this patient population. | 2 years

SECONDARY OUTCOMES:
To make a preliminary assessment of the anti-tumor activity of these combinations. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Peter C. Enzinger, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts